CLINICAL TRIAL: NCT03148275
Title: A Non-Randomized, Open-Label, Phase 2 Study of Trametinib in Patients With Unresectable or Metastatic Epithelioid Hemangioendothelioma
Brief Title: Trametinib in Treating Patients With Epithelioid Hemangioendothelioma That is Metastatic, Locally Advanced, or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00712; NCI-2017-00712 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SARC033; 10015 (Other: University of Michigan Comprehensive Cancer Center EDDOP); 10015 (Other: CTEP); P30CA046592 (NIH)
Record Dates: First submitted 2017-05-01; First posted 2017-05-10 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Locally Advanced Epithelioid Hemangioendothelioma; Metastatic Epithelioid Hemangioendothelioma; Unresectable Epithelioid Hemangioendothelioma
MeSH Terms: conditions — Hemangioendothelioma, Epithelioid | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trametinib) (Experimental): Patients receive trametinib PO QD on days 1-28. Treatment repeats every 28 days for up to 52 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Drug: Trametinib

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK-1120212; GSK1120212; JTP-74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase II trial studies how well trametinib works in treating patients with epithelioid hemangioendothelioma that has spread to other places in the body (metastatic), nearby tissue or lymph nodes (locally advanced), or cannot be removed by surgery (unresectable). Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimate the objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

SECONDARY OBJECTIVES:

I. Estimate the 6-month and median progression free survival (PFS) rates. II. Estimate the 2-year and median overall survival (OS) rates. III. Evaluate the safety of trametinib in patients with epithelioid hemangioendothelioma.

IV. Evaluate patient-reported symptoms using National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) global health; pain intensity, interference and behavior short form inventories prior to, after 4 weeks and after 6 months (if stable or better disease) of treatment, and on evidence of disease progression.

EXPLORATORY OBJECTIVES:

I. Compare the rates of epithelioid hemangioendothelioma progression prior to starting trametinib to rates on treatment by central review of radiology images.

II. Evaluate the effect of trametinib on change in tumor volume and compare to RECIST 1.1 response through central imaging review.

III. Evaluate the effect of trametinib on markers of inflammation including c-reactive protein (CRP), erythrocyte sedimentation rate (ESR) and plasma connective tissue growth factor (CTGF).

OUTLINE:

Patients receive trametinib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 52 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam; baseline imaging must be obtained within 30 days of day 1 of study
* Patients must have histologically confirmed epithelioid hemangioendothelioma which is metastatic or locally advanced (unresectable), and tumor tissue (paraffin-embedded tissue block or tumor tissue on unstained glass slides) available for fusion fluorescence in situ hybridization (FISH) analysis at Cleveland Clinic; patient tumor tissue stored in pathology archives may be used for fusion FISH; a new biopsy is not mandatory
* Patients must have evidence of disease progression per RECIST 1.1 prior to enrollment or have evidence of cancer-related pain requiring symptom management with narcotic analgesics
* Because there is no established standard or approved drug therapy for treatment of epithelioid hemangioendothelioma (EHE), patients previously untreated or treated with drug therapy for EHE are eligible; there is no limit on the number of prior regimens used to be eligible
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Able to swallow orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or small bowel
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5) grade =< 1 (except alopecia) at the time of enrollment
* Absolute neutrophil count (ANC) >= 1 x 10^9/L (within 2 weeks of patient registration)
* Hemoglobin >= 9 g/dL, patients may receive transfusion to meet criterion (within 2 weeks of patient registration)
* Platelets >= 75 x 10^9/L (within 2 weeks of patient registration)
* Albumin >= 2.5 g/dL (within 2 weeks of patient registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 2 weeks of patient registration); NOTE: patients with elevated bilirubin secondary to Gilbert's disease are eligible to participate in the study
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN (within 2 weeks of patient registration)
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min (within 2 weeks of patient registration)
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) or multigated acquisition scan (MUGA) (within 30 days of registration)
* Trametinib can cause fetal harm when administered to a pregnant woman; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for four months after the last dose of the drug; women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to enrollment and agree to use effective contraception throughout the treatment period and for 4 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Human immunodeficiency virus (HIV)-patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, however HIV-positive patients must meet the following criteria:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based test

Exclusion Criteria:

* Prior systemic therapy with a MEK inhibitor
* History of another malignancy

  * Exception: patients who have been disease-free for 3 years or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies, are eligible; consult the Cancer Therapy Evaluation Program (CTEP) medical monitor if unsure whether second malignancies meet the requirements specified above
* History of interstitial lung disease or pneumonitis requiring supplemental oxygen or treatment with oral or intravenously administered corticosteroids
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity (e.g. doxorubicin), biologic therapy, or immunotherapy within 21 days prior to enrollment and/or daily or weekly chemotherapy (e.g. sunitinib, sorafenib and pazopanib) without the potential for delayed toxicity within 14 days prior to enrollment
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of trametinib and during the study
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients or to dimethyl sulfoxide (DMSO)
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * Because the composition, pharmacokinetics (PK), and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* History or current evidence/risk of retinal vein occlusion (RVO)
* History or evidence of cardiovascular risk including any of the following:

  * A QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators
  * Known cardiac metastases
* Known hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible)
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Trametinib was embryotoxic and abortifacient in rabbits at doses greater than or equal to those resulting in exposures approximately 0.3 times the human exposure at the recommended clinical dose. Therefore, the study drug must not be administered to pregnant women or nursing mothers; women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; if a female patient or a female partner of a patient becomes pregnant while the patient receives trametinib, the potential hazard to the fetus should be explained to the patient and partner (as applicable)
* Inability to comply with protocol-required procedures

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Schuetze, Principal Investigator — University of Michigan Comprehensive Cancer Center EDDOP
Locations (36):
- United States (36):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Ma S, Kanai R, Pobbati AV, Li S, Che K, Seavey CN, Hallett A, Burtscher A, Lamar JM, Rubin BP. The TAZ-CAMTA1 Fusion Protein Promotes Tumorigenesis via Connective Tissue Growth Factor and Ras-MAPK Signaling in Epithelioid Hemangioendothelioma. Clin Cancer Res. 2022 Jul 15;28(14):3116-3126. doi: 10.1158/1078-0432.CCR-22-0421. PMID 35443056

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Trametinib): Patients received trametinib PO QD on days 1-28. Treatment repeats every 28 days for up to 52 cycles in the absence of disease progression or unacceptable toxicity.
  Questionnaire Administration: Ancillary studies
  Trametinib: Given PO
Period: Overall Study
Arm/Group | Treatment (Trametinib)
Started | 44
Completed | 25
Not Completed | 19
Not completed — Death | 6
Not completed — Adverse Event | 3
Not completed — Liver transplant | 2
Not completed — Patient decision | 5
Not completed — transition to commercial drug | 1
Not completed — subjects withdrew from the trial after registration, but before starting study treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 54 [22 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1. A Simon minimax sampling two-stage design will be used to estimate the objective response rate. Will be calculated along with 95% confidence intervals.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 42
Percentage | 9.5 [3.1 to 23.5]

2. Secondary Outcome: 6 Month Progression-free Survival
Description: Will be calculated along with 95% confidence intervals and estimated by the Kaplan-Meier method.
Time Frame: From time of first dose of study medication to occurrence of radiologic tumor progression per Response Evaluation Criteria in Solid Tumors 1.1, clinical progression based on treating physician assessment or death from any cause, assessed at 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 42
percentage of participants | 66.5 [53.6 to 82.5]

3. Secondary Outcome: Overall Survival
Description: Will be calculated along with 95% confidence intervals and estimated by the Kaplan-Meier method.
Time Frame: From the time of first dose of study drug to occurrence of death from any cause, assessed at 2 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 42
Percentage | 41.1 [28.1 to 60.1]

4. Secondary Outcome: Incidence of Adverse Events
Description: Graded according to the National Cancer Institute Common Terminology Criteria of Adverse Events version 5.0. The rates of adverse events occurring in at least 5% of subjects and rates of grade 3-5 adverse events will be tabulated by system and term.
Time Frame: at 6 months
Measure: Number; unit: participants who experienced the event
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 42
participants who experienced the event
  Abdominal Pain | 3
  Alanine Aminotransferase Increased | 8
  Alkaline Phosphatase Increased | 8
  Alopecia | 13
  Anemia | 21
  Anorexia | 11
  Anxiety | 6
  Aspartate Aminotransferase Increased | 13
  Blurred Vision | 6
  Bruising | 3
  Constipation | 18
  Cough | 9
  Creatinine Increased | 6
  Dehydration | 8
  Diarrhea | 22
  Dizziness | 12
  Dry Mouth | 6
  Dry Skin | 9
  Dysgeusia | 4
  Dyspnea | 20
  Edema Face | 4
  Edema Limbs | 21
  Fatigue | 28
  Fever | 5
  Headache | 3
  Hyperglycemia | 6
  Hypertension | 15
  Hypoalbuminemia | 19
  Hypocalcemia | 11
  Hypokalemia | 6
  Hyponatremia | 10
  Hypotension | 7
  Hypoxia | 7
  Lymphocyte Count Decreased | 7
  Mucositis Oral | 8
  Myalgia | 3
  Nausea | 24
  Neutrophil Count Decreased | 6
  Non-Cardiac Chest Pain- Grade 1 | 7
  Oral Pain | 3
  Pain | 8
  Pain In Extremity | 9
  Palpitations | 5
  Paresthesia | 4
  Paronychia | 4
  Platelet Count Decreased | 7
  Pleural Effusion | 7
  Productive Cough | 3
  Pruritus | 9
  Rash Acneiform | 21
  Rash Maculo-Papular | 13
  Sinus Tachycardia | 4
  Skin Infection | 6
  Sore Throat | 4
  Syncope | 4
  Upper Respiratory Infection | 4
  Urinary Tract Infection | 4
  Vomiting | 18
  Weight Gain | 5
  Back Pain | 4
  Fall | 3
  Hyperkalemia | 5
  Insomnia | 4
  Neck pain | 3
  Respiratory failure | 4
  Skin ulceration | 3
  Weight loss | 7
  White blood cell decreased | 4
  Acute kidney injury- Grade 3 | 1
  Agitation- Grade 3 | 1
  Alanine aminotransferase increased- Grade 3 | 1
  Alkaline phosphatase increased- Grade 3 | 2
  Altered mental status- Grade 3 | 1
  ammonia high- Grade 3 | 1
  Anemia- Grade 3 | 6
  Anxiety- Grade 3 | 2
  Aspartate aminotransferase increased- Grade 3 | 3
  Aspiration- Grade 3 | 1
  Back Pain- Grade 3 | 1
  Bullous dermatitis- Grade 3 | 1
  Cellulitis- Grade 3 | 1
  Chest wall pain- Grade 3 | 2
  Cholecystitis- Grade 3 | 1
  Colitis- Grade 3 | 2
  Confusion- Grade 3 | 1
  Constipation- Grade 3 | 1
  Duodenal hemorrhage- Grade 3 | 1
  Dysesthesia- Grade 3 | 1
  Dysphagia- Grade 3 | 1
  Dyspnea- Grade 3 | 3
  Edema Limbs- Grade 3 | 1
  Encephalopathy- Grade 3 | 1
  Fatigue- Grade 3 | 2
  Flank Pain- Grade 3 | 1
  Gamma-glutamyl transferase- Grade 3 | 1
  Gastric hemorrhage- Grade 3 | 1
  Heart Failure- Grade 3 | 1
  Hemoptysis- Grade 3 | 1
  Hepatic failure- Grade 3 | 1
  Hyperglycemia- Grade 3 | 1
  Hyperkalemia- Grade 3 | 1
  Hypertension- Grade 3 | 4
  Hypoalbuminemia- Grade 3 | 2
  Hypoglycemia- Grade 3 | 1
  Hyponatremia- Grade 3 | 3
  Hypotension- Grade 3 | 3
  Hypoxia- Grade 3 | 3
  Liver transplant- Grade 3 | 1
  Lung infection- Grade 3 | 2
  melena- Grade 3 | 1
  Mucositis oral- Grade 3 | 1
  Pleural effusion- Grade 3 | 2
  Pleural infection- Grade 3 | 1
  Pneumonitis- Grade 3 | 1
  Portal vein thrombosis- Grade 3 | 2
  Pulmonary hypertension- Grade 3 | 1
  Rash acneiform- Grade 3 | 3
  Rash maculo-papular- Grade 3 | 1
  Respiratory failure- Grade 3 | 1
  Skin infection- Grade 3 | 1
  Supraventricular tachycardia- Grade 3 | 1
  Syncope- Grade 3 | 3
  Tumor Pain- Grade 3 | 1
  Urinary tract infection- Grade 3 | 1
  Urine output decrease- Grade 3 | 1
  weight loss- Grade 3 | 1
  Hypokalemia- Grade 4 | 1
  Obesity- Grade 4 | 1
  Platelet count decreased- Grade 4 | 1
  Respiratory failure- Grade 4 | 2
  Adult respiratory distress- Grade 5 | 1
  Cardiac arrest- Grade 5 | 1
  Death NOS- Grade 5 | 6
  Duodenal hemorrhage- Grade 5 | 1
  Respiratory failure- Grade 5 | 2
  Stridor- Grade 5 | 1
  Upper gastrointestinal hemorrhage- Grade 5 | 1

5. Secondary Outcome: Change in Patient Reported Symptoms
Description: Will be assessed by the National Institutes of Health Patient Reported Outcomes Measurement Information System questionnaire. Patient Reported Outcomes Measurement Information System questionnaires will be scored according to recommended standardized system and t-scores generated. A mixed model will be used to analyze change in t-scores over time. PROMIS questionnaires were scored according to recommended standardized system and T-scores. A Wilcoxon signed rank test was used to assess the change in scores/T-scores over time. Determination of change in score between timepoints only included patients that had scores at those timepoints.
  Pain Intensity - 3a Scale: 36.3 (no pain) - 81.8 (severe pain) Pain Interference - 4a Scale: 41.6 (no interference) - 75.6 (large interference) Pain Behavior - 7a Scale: 34.1 (had no pain) - 78.9 (always in pain) Global Mental Heath Scale: 21.2 (severe) - 67.6 (none) Global Mental Physical Scale: 16.2 (severe) - 67.7 (none)
Time Frame: Baseline and at 6 months
Population: as participants were removed from trial, the number of completed PROMIS forms decreased
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 42
T Score
  Pain Intensity - 3a: Baseline | 57 (12)
  Pain Intensity - 3a: 4 weeks: number analyzed (Participants) | 36
  Pain Intensity - 3a: 4 weeks | 52 (11)
  Pain Intensity - 3a: 6 months: number analyzed (Participants) | 20
  Pain Intensity - 3a: 6 months | 49 (11)
  Pain Interference - 4a: Baseline | 59 (11)
  Pain Interference - 4a: 4 weeks: number analyzed (Participants) | 36
  Pain Interference - 4a: 4 weeks | 54 (11)
  Pain Interference - 4a: 6 months: number analyzed (Participants) | 20
  Pain Interference - 4a: 6 months | 51 (9)
  Pain Behavior - 7a: Baseline: number analyzed (Participants) | 39
  Pain Behavior - 7a: Baseline | 56 (11)
  Pain Behavior - 7a: 4 weeks: number analyzed (Participants) | 35
  Pain Behavior - 7a: 4 weeks | 53 (11)
  Pain Behavior - 7a: 6 months: number analyzed (Participants) | 20
  Pain Behavior - 7a: 6 months | 51 (12)
  Global Mental Heath (questions 2,4,5,10): Baseline | 43 (10)
  Global Mental Heath (questions 2,4,5,10): 4 weeks: number analyzed (Participants) | 37
  Global Mental Heath (questions 2,4,5,10): 4 weeks | 42 (8)
  Global Mental Heath (questions 2,4,5,10): 6 months: number analyzed (Participants) | 20
  Global Mental Heath (questions 2,4,5,10): 6 months | 38 (10)
  Global Physical Health (questions 3,6,7,8): Baseline | 41 (10)
  Global Physical Health (questions 3,6,7,8): 4 weeks: number analyzed (Participants) | 37
  Global Physical Health (questions 3,6,7,8): 4 weeks | 36 (8)
  Global Physical Health (questions 3,6,7,8): 6 months: number analyzed (Participants) | 20
  Global Physical Health (questions 3,6,7,8): 6 months | 36 (9)

6. Secondary Outcome: Median Progression-free Survival
Description: Will be calculated along with 95% confidence intervals and estimated by the Kaplan-Meier method.
Time Frame: From time of first dose of study medication to occurrence of radiologic tumor progression per Response Evaluation Criteria in Solid Tumors 1.1, clinical progression based on treating physician
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 42
months | 8.3 [7.3 to 21.9]

7. Other Pre Specified Outcome: Change in Epithelioid Hemangioendothelioma Growth Rate
Description: McNemar test will be used to compare the number of patients with epithelioid hemangioendothelioma progression prior to starting trametinib to the number of patients with epithelioid hemangioendothelioma progression during treatment.
Time Frame: Baseline up to 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in CRP Level
Description: Will be used as time-dependent variables in a Cox model to determine the association with epithelioid hemangioendothelioma survival.
Time Frame: Baseline up to 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in ESR Level
Description: as for outcome 8
Time Frame: Baseline up to 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Plasma CTGF Level
Description: Will be analyzed by enzyme-linked immunosorbent assay. Will be used as time-dependent variables in a Cox model to determine the association with epithelioid hemangioendothelioma survival.
Time Frame: Baseline up to 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Tumor Volume
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1. Will be summarized with a scatterplot. The Pearson correlation coefficient (or Spearman, if more appropriate) will be assessed to determine the strength of the agreement. Agreement of the tumor classifications (response versus no response) will be summarized as the raw agreement and with a Kappa Statistic. The association of the change in tumor volume with survival will be evaluated in two ways. The first will be to use the change in tumor volume as a time dependent variable in a Cox model. The second will be a landmark analysis (done at either the first radiographic assessment or at the second radiographic assessment) to compare the survival of patients classified as a responder (based on tumor volume) to those who have not responded by the selected landmark time. Patients who died prior to the landmark time point will be omitted from analysis.
Time Frame: Baseline up to 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of TAZ-CAMTA1 Gene Fusion
Description: Will be evaluated by fluorescence in situ hybridization.
Time Frame: Up to 6 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Percent of TAZ-CAMTA1 Gene Fusion
Description: Will be evaluated by fluorescence in situ hybridization.
Time Frame: Up to 6 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: MAP Kinase Activation
Description: Will be analyzed by immunohistochemistry. Descriptive statistics will be generated, and estimates for the proportion of samples with demonstrated inhibition of MAPK signaling post-treatment compared to pre-treatment will be generated along with 95% confidence intervals. Likewise, the proportion of patients with demonstrated MAPK signaling inhibition at time of disease progression will be determined with the corresponding 95% confidence interval.
Time Frame: Up to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: data was collected over 6 years
Arm/Group | Treatment (Trametinib)
All-Cause Mortality (participants affected / at risk) | 27/42
Serious Adverse Events (participants affected / at risk) | 25/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trametinib) (N=42)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Altered mental status (Psychiatric disorders) | 1 (1)
Anemia (Investigations) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Bullous dermatitis (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
cellulitis (Infections and infestations) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Dysesthesia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema limbs (General disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flank pain (General disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Liver Transplant (Renal and urinary disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural infection (Infections and infestations) | 1 (1)
Pneumonitis (Infections and infestations) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trametinib) (N=42)
Abdominal pain (Gastrointestinal disorders) | 3 (10)
Alanine aminotransferase increased (Investigations) | 8 (15)
Alkaline phosphatase increased (Investigations) | 8 (28)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13)
Anemia (Investigations) | 21 (62)
Anorexia (Metabolism and nutrition disorders) | 11 (15)
Anxiety (Psychiatric disorders) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 13 (35)
Blurred vision (Eye disorders) | 6 (9)
Bruising (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 18 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Creatinine increased (Investigations) | 6 (14)
Dehydration (Metabolism and nutrition disorders) | 8 (11)
Diarrhea (Gastrointestinal disorders) | 22 (43)
Dizziness (General disorders) | 12 (21)
Dry mouth (General disorders) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9)
Dysgeusia (General disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 (27)
Edema face (General disorders) | 4 (4)
Edema limbs (General disorders) | 21 (38)
Fatigue (General disorders) | 28 (42)
Fever (General disorders) | 5 (6)
Headache (General disorders) | 3 (4)
Hyperglycemia (Investigations) | 6 (14)
Hypertension (Vascular disorders) | 15 (24)
Hypoalbuminemia (Investigations) | 19 (47)
Hypocalcemia (Investigations) | 11 (16)
Hypokalemia (Investigations) | 6 (10)
Hyponatremia (Investigations) | 10 (16)
Hypotension (Vascular disorders) | 7 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Lymphocyte count decreased (Investigations) | 7 (10)
Mucositis oral (General disorders) | 8 (12)
Myalgia (General disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 24 (35)
Neutrophil count decreased (Investigations) | 6 (9)
Non-cardiac chest pain (General disorders) | 7 (10)
Oral pain (General disorders) | 3 (6)
Pain (General disorders) | 8 (11)
Pain in extremity (General disorders) | 9 (10)
Palpitations (Vascular disorders) | 5 (5)
Paresthesia (General disorders) | 4 (4)
Paronychia (Infections and infestations) | 4 (9)
Platelet count decreased (Investigations) | 7 (13)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 21 (51)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (23)
Sinus tachycardia (Vascular disorders) | 4 (4)
Skin infection (Infections and infestations) | 6 (9)
Sore throat (General disorders) | 4 (4)
Syncope (Nervous system disorders) | 4 (4)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Urinary tract infection (Infections and infestations) | 4 (6)
Vomiting (Gastrointestinal disorders) | 18 (31)
Weight gain (General disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Fall (General disorders) | 3 (3)
Hyperkalemia (Investigations) | 5 (7)
Insomnia (Psychiatric disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (5)
Weight loss (General disorders) | 7 (14)
White blood cell decreased (Investigations) | 4 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT03148275/Prot_SAP_000.pdf